CLINICAL TRIAL: NCT07277010
Title: Building an Artificial Intelligence-Driven Early Warning System and Home Management Protocol for a Diabetic Foot Ulcer Recurrence Cohort
Brief Title: AI Wound Alert & Home Management for Recurrent DFU
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Long Zhang, Head of Wound Healing Center, Peking University Third Hospital
Other Study IDs: Long2025-DFU-recurrence cohort
Record Dates: First submitted 2025-11-30; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Diabetic Foot Ulcer (DFU)
Keywords: diabetic foot ulcer; recurrent; precaution
MeSH Terms: conditions — Diabetic Foot; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The population with DFU recovery: The wound was caused by diabetic foot. After treatment, the wound healed. The healing criteria were as follows: the wound was dry with no exudate; the wound bed and edges were completely epithelialized; there were no signs of redness or swelling in the surrounding area; and the wound had sufficient tensile strength to withstand pressure without cracking
  Interventions: Behavioral: Individualized follow-up care

INTERVENTIONS:
Behavioral: Individualized follow-up care — Re-classification system for high-risk feet, along with individualized follow-up care

SUMMARY:
Diabetes is one of the major chronic diseases, and diabetic foot ulcer (DFU) is a significant adverse prognosis of diabetes. The recurrence of DFU after healing involves multiple risk factors, such as changes in foot loading patterns, patient compliance, family care capacity, blood glucose monitoring, the degree of ischemia, and control of systemic diseases. Early identification of signs of DFU recurrence and timely follow-up interventions are crucial for improving prognosis, reducing disability rates, and lowering healthcare costs. However, traditional follow-up systems lack individualized strategies (e.g., insufficient risk stratification, rigid follow-up intervals, inadequate compliance management), often resulting in low follow-up efficacy. High-risk patients prone to recurrence may not receive frequent enough follow-ups for early detection, while low-risk patients unlikely to recur may undergo multiple unnecessary visits, increasing the burden on both patients and healthcare providers. This inefficiency is a key reason for the persistently high rates of disability and mortality among patients with recurrent DFU. Establishing individualized follow-up strategies for DFU, leveraging advanced technologies to address core bottlenecks such as delayed recurrence warnings and insufficient home management, represents an effective technical approach to solving these problems.

Our center aims to establish and refine a specialized cohort for active DFU follow-up, along with a multimodal database with comprehensive indicators. We plan to explore a high-risk foot grading system for preventing DFU recurrence and develop targeted follow-up protocols. Using AI technology, we will create a wound alert system capable of identifying DFU recurrence and explore a remote healthcare and AI-assisted prevention and control system for DFU recurrence, centered on patient self-management at home.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of type 1 or type 2 diabetes in accordance with the definitions set by the World Health Organization；
* The wound was caused by diabetic foot*. After treatment, the wound healed. The criteria for successful healing were as follows: the wound was dry with no exudate; the wound bed and edges were completely epithelialized; there were no signs of redness or swelling in the surrounding area; and the wound had sufficient tensile strength to withstand pressure without cracking；
* Voluntarily participated in this study and signed the informed consent form.

Exclusion Criteria:

* The patient is unable to cooperate or has a mental disorder；
* At the discretion of the researchers, the subject is not suitable for this study or is unable to comply with the requirements of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population with DFU recovery
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
1-year recurrence rate of diabetic foot | 1-year
  Recurrence rate of diabetic foot = (Number of diabetic foot patients who experience ulcer recurrence within 1 year) / (Total number of diabetic foot patients whose ulcers have healed) × 100%

SECONDARY OUTCOMES:
Proportion of patients with Wagner grade 1/2 among those who experienced DFU recurrence within 1 year of follow-up | 1-year
  Number of patients with Wagner stage 1/2 among those who experienced DFU recurrence within 1 year of follow-up / Total number of patients who experienced DFU recurrence within 1 year of follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided